CLINICAL TRIAL: NCT02235909
Title: A Randomized, Double-Blind, Efficacy and Safety Study of AR 14 (AZILSARTAN MEDOXOMIL) Treatment and Withdrawal, Followed by an Open-Label Extension, in Children 6 to Less Than 18 Years of Age With Hypertension
Brief Title: An Efficacy and Safety Study in Children 6 to Less Than 18 Years of Age With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR14.001
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: Pediatric Hypertension; High Blood Pressure; Hypertension; Pediatric; Primary Hypertension; Secondary Hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — azilsartan medoxomil; Losartan

STUDY DESIGN:
Intervention Model Description: There are 3 phases in this study. Double-blind, withdrawal phase, and open-label phase.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind masking in the Double Blind Phase and Withdrawal Phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Double-blind: Azilsartan Medoxomil - Low dose (Experimental): 6-week, double-blind (DB), randomized, treatment phase (DB Phase): Azilsartan medoxomil low-dose (AZM-L), 10 mg once daily.
  Interventions: Drug: Azilsartan Medoxomil Low-dose
- Double blind phase: Losartan (Active Comparator): 6-week, double-blind (DB), randomized, treatment phase (DB Phase): Starting at Losartan 25/50 and force titrated to 50/100 mg daily at Week 2.
  Interventions: Drug: Losartan
- Withdrawal Phase: Azilsartan medoxomil low-dose (AZM-L) (Active Comparator): Experimental Arm in the Withdrawal Phase, subjects will be randomized (1:1) to continue taking their previously assigned active treatment (AZM-L) that was taken in Double blind OR to be switched to placebo.
  Interventions: Drug: Azilsartan Medoxomil Low-dose
- Withdrawal Phase: Placebo to match azilsartan medoxomil low dose (AZM-L) (Placebo Comparator): Placebo Arm in the Withdrawal Phase for subjects who were on AZM-L in double blind then randomized (1:1) to placebo for withdrawal phase
  Interventions: Drug: Losartan
- Open Label Phase: Azilsartan Medoxomil (Experimental): Azilsartan Medoxomil 10 mg which can be titrated to higher dose(s) (up to 40 mg for subjects <50 kg or up to 80 mg for subjects ≥50 kg)
  Interventions: Drug: Azilsartan Medoxomil Low-dose
- Withdrawal Phase: Losartan 50 mg (Active Comparator): Withdrawal Phase, subjects will be randomized (1:1) to continue taking their previously assigned active treatment or to be switched to placebo.
  Interventions: Drug: Losartan
- Withdrawal Phase: Placebo to Losartan (Placebo Comparator): Placebo Arm In the Withdrawal Phase, subjects will be randomized (1:1) to continue taking their previously assigned active treatment or to be switched to placebo.
  Interventions: Drug: Placebo for Losartan
- Double-blind: Azilsartan Medoxomil - Medium dose (Experimental): 6-week, double-blind (DB), randomized, treatment phase (DB Phase), Azilsartan medoxomil Medium-dose (AZM-M), 20 mg once daily at Week 2.
  Interventions: Drug: Azilsartan Medoxomil Low-dose; Drug: Placebo for Losartan; Drug: Azilsartan Medoxomil Medium-dose (20 mg)
- Double-blind: Azilsartan Medoxomil - High dose (AZM-H) (Experimental): 6-week, double-blind (DB), randomized, treatment phase (DB Phase): Azilsartan medoxomil High-dose (AZM-H), 40 mg AZM-M
  Interventions: Drug: Azilsartan Medoxomil High-dose (40 mg)
- Withdrawal: Azilsartan Medoxomil - Medium dose (Experimental): Experimental Arm in the Withdrawal Phase, subjects will be randomized (1:1) to continue taking their previously assigned active treatment (AZM-M) that was taken in Double blind OR to be switched to placebo.
  Interventions: Drug: Azilsartan Medoxomil Low-dose; Drug: Azilsartan Medoxomil Medium-dose (20 mg)
- Withdrawal: Azilsartan Medoxomil - High dose (Experimental): Experimental Arm in the Withdrawal Phase, subjects will be randomized (1:1) to continue taking their previously assigned active treatment (AZM-H) that was taken in double blind OR to be switched to placebo.
  Interventions: Drug: Azilsartan Medoxomil High-dose (40 mg)
- Withdrawal Phase: Placebo to match azilsartan medoxomil medium dose (AZM-M) (Experimental): Placebo arm in the Withdrawal Phase for subjects who were on AZM-M in double blind then randomized (1:1) to matching placebo for withdrawal phase
  Interventions: Drug: Placebo for Azilsartan Medoxomil
- Withdrawal Phase: Placebo to match azilsartan medoxomil high dose (AZM-H) (Experimental): Placebo arm in the Withdrawal Phase for subjects who were on AZM-H in Double blind then randomized (1:1) to matching placebo for withdrawal phase
  Interventions: Drug: Placebo for Azilsartan Medoxomil

INTERVENTIONS:
Drug: Azilsartan Medoxomil Low-dose — Azilsartan medoxomil low-dose (AZM-L) 10 mg
  Other Names: AR14; AZM-L
  Arms: Double-blind: Azilsartan Medoxomil - Low dose; Double-blind: Azilsartan Medoxomil - Medium dose; Open Label Phase: Azilsartan Medoxomil; Withdrawal Phase: Azilsartan medoxomil low-dose (AZM-L); Withdrawal: Azilsartan Medoxomil - Medium dose
Drug: Losartan
  Other Names: Cozaar
  Arms: Double blind phase: Losartan; Withdrawal Phase: Losartan 50 mg; Withdrawal Phase: Placebo to match azilsartan medoxomil low dose (AZM-L)
Drug: Placebo for Azilsartan Medoxomil
  Arms: Withdrawal Phase: Placebo to match azilsartan medoxomil high dose (AZM-H); Withdrawal Phase: Placebo to match azilsartan medoxomil medium dose (AZM-M)
Drug: Placebo for Losartan
  Arms: Double-blind: Azilsartan Medoxomil - Medium dose; Withdrawal Phase: Placebo to Losartan
Drug: Azilsartan Medoxomil Medium-dose (20 mg) — Azilsartan medoxomil medium-dose (AZM-M) 20 mg
  Other Names: AR14; AZM-M
  Arms: Double-blind: Azilsartan Medoxomil - Medium dose; Withdrawal: Azilsartan Medoxomil - Medium dose
Drug: Azilsartan Medoxomil High-dose (40 mg) — Azilsartan medoxomil high-dose (AZM-L) 40 mg
  Other Names: AR14; AZM-H
  Arms: Double-blind: Azilsartan Medoxomil - High dose (AZM-H); Withdrawal: Azilsartan Medoxomil - High dose

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of the study drug relative to an active comparator losartan which is in the same class of drug and is approved for use in the pediatric population aged 6 years and older. Approximately 260 subjects will participate in a 6-week, double-blind, randomized, treatment phase, followed by a 2-week, double-blind, randomized, placebo-controlled withdrawal phase. A 44-week, open-label extension in which all subjects will receive azilsartan and other antihypertensive medications (if needed). Blood pressure will be assessed throughout the study.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy and safety of the study drug relative to an active comparator losartan which the same class of drug and is approved for use in the pediatric population aged 6 years and older. Approximately 260 subjects will participate in a 6-week, double-blind, randomized, treatment phase, followed by a 2-week, double-blind, randomized, placebo-controlled withdrawal phase. This study also includes a 44-week, open-label extension Phase in which all subjects will receive azilsartan and other antihypertensive medications (if needed) in order to reach an optimal blood pressure. Blood pressure will be assessed in the clinic throughout the study, and subjects may also participate in a 24-hour ambulatory blood pressure monitoring procedure at baseline, at the end of the double-blind Phase and at the end of the open-label Phase.

ELIGIBILITY:
Inclusion Criteria:

* The subject has hypertension (primary or secondary) defined as clinic Seated Diastolic BP ≥95th percentile (by age, gender, and height) or ≥90th percentile (by age, gender, height) if chronic renal disease, diabetes, heart failure or hypertensive target organ damage is present

  1. If currently treated: The subject has a documented historical diagnosis of hypertension AND a post-washout clinic Seated Diastolic BP meeting the above criteria on Day -1 (or Day 1 for subjects not participating in Ambulatory Blood Pressure Monitoring)
  2. If currently untreated: The subject has elevated Seated Diastolic BP meeting the above criteria on 3 separate occasions before Randomization, including on Day -1 (or Day 1 for subjects not participating in Ambulatory Blood Pressure Monitoring)
* The subject is male or female and aged 6 to <18 years at Baseline and weighs at least 25 kg
* The subject agrees to continue their previously implemented nonpharmacological life style modifications if begun prior to Screening. Note: For subjects participating in a weight loss program, the weight maintenance

Exclusion Criteria:

* The subject has a clinic Seated Diastolic BP greater than 15 mm Hg and/or Seated Diastolic BP greater than 10 mm Hg above the 99th percentile for age, gender, and height as confirmed by the average (arithmetic mean) of 3 serial clinic seated BP measurements at Screening/Visit 1
* The subject has a diagnosis of malignant or accelerated hypertension
* The subject is currently treated with more than 2 antihypertensive agents
* The subject or parent/legal guardian is not willing for the subject's previous antihypertensive medications to be stopped
* The subject has participated in the intensive, active weight-loss phase of a weight-loss program within 30 days prior to Screening/Visit 1
* The subject has any of the following: severe renal impairment (eGFR <30 mL/min/1.73 m2 by the Schwartz formula); is currently undergoing dialysis treatment; renovascular disease affecting both kidneys or a solitary kidney; severe nephrotic syndrome not in remission; or serum albumin <2.5 g/dL
* The subject has a history or clinical manifestations of severe cardiovascular, hepato-biliary, gastrointestinal, endocrine-metabolic (e.g., hyperthyroidism, Cushing's syndrome), hematologic, immunologic, genito-urinary, or psychiatric disease, cancer, and/or any conditions that would interfere with the health status of the subject through study participation, or would jeopardize study integrity in the opinion of the investigator
* The subject is suffering from uncorrected coarctation of the aorta, or hemodynamically significant left ventricular outflow tract obstruction due to eg, aortic valvular disease, or is likely to undergo a procedure known to affect blood pressure (eg, repair of arterial anomalies) during the course of the study
* The subject is poorly controlled diabetic defined as having a glycosylated hemoglobin value >8.5% at Screening/Visit 1
* The subject has hyperkalemia as defined by the central laboratory's normal reference range or any pertinent electrolyte disorders at Screening/Visit

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 377 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Caras, MD, Study Director — Arbor Pharmaceuticals, LLC
Locations (69):
- United States (17):
  - Advanced Research Center, INC, Anaheim, California
  - Direct Helpers Research Center, Hialeah, Florida
  - JDH Medical Group LLC, Miami, Florida
  - University of Miami/Jackson Memorial Hospital, Miami, Florida
  - Medical Research Center of Miami II, Inc., Miami, Florida
  - Pioneer Clinical Research, North Miami, Florida
  - Georgia Clinical Research, Snellville, Georgia
  - Zoe Center for Pediatrics, Thomaston, Georgia
  - University of Louisville, Louisville, Kentucky
  - David M. Headley, MD PA, Port Gibson, Mississippi
  - Mount Sinai PRIME, Lake Success, New York
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Memphis and Shelby County Pediatric Group, Memphis, Tennessee
  - Southeast Texas Clinical Research Center, Beaumont, Texas
  - Texas Children's Heart Center, Houston, Texas
  - Ericksen Research & Development, LLC, Clinton, Utah
  - Mid-Columbia Research, Richland, Washington
- Argentina (3):
  - Hospital Italiano, Ciudad Autonoma, Buenos Aires
  - Hospital de Niños, Ciudad Autonoma, Buenos Aires
  - Clinica de Nefrologia, Urologia y Enf. Cardiovasculares S A, Santa Fe
- Brazil (6):
  - Clínica Nefrokids Ltda, Curitiba
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre
  - Fundação José Luiz Egydio Setúbal, São Paulo
  - Hospital Samaritano, São Paulo
  - Eurolatino Pesquisas Médicas Ltda., Uberlândia
- SHATPPD-Ruse EOOD, Rousse, Bulgaria
- Colombia (5):
  - Fundacion Oftalmologica de Santander - FOSCAL, Bucaramanga
  - Fundacion Valle del Lili, Cali
  - Fundacion Hospitalaria San Vicente de Paul, Medellín
  - Hospital Pablo Tobón Uribe, Medellín
  - Institucion Prestadora de Servicios de Salud de la Universidad de Antioquia "IPS UNIVERSITARIA", Medellín
- Hungary (5):
  - Principal SMO Kft., Baja
  - Svabhegy Plusz Gyermekegeszsegugyi Kozpont, Budapest
  - Szent Lukacs Korhaz Dombovar, Dombóvár
  - Prehospital Med Kft., Miskolc
  - Szegedi Tud.Egyetem Szent-Gyorgyi Albert Klin. Kozp., Szeged
- Italy (3):
  - Ospedale Pediatrico Giovanni XXIII, Bari
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - A.R.N.A.S. Ospedale Civico e Benfratelli, G. Cristina e M.Ascoli, Palermo
- Mexico (4):
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Hospital General de Mexico, Mexico City
  - Accelerium S. de R.L. de C.V., Monterrey
  - Centro de Investigacion Clinica Chapultepec S.A. de C.V., Morelia
- Poland (4):
  - SPZOZ Uniwersytecki Dzieciecy Szpital Kliniczny im. L. Zamenhofa, Bialystok
  - Uniwersytecki Szpital Dziecięcy w Krakowie, Krakow
  - NZOZ TRI-medica, Lodz
  - Praktyka Lekarzy Rodzinnych R.Jadach, M.Domanski NZOZ, Wroclaw
- South Africa (6):
  - LCS Clinical Research Unit, Johannesburg, Gauteng
  - Soweto Clinical Trial Centre, Soweto, Gauteng
  - Netcare St. Anne's Hospital, Pietermaritzburg, KwaZulu-Natal
  - Groote Schuur Hospital E13 Renal Unit, Cape Town, Western Cape
  - Clinical Projects Research SA (PTY) LTD, Worcester, Western Cape
  - CRISMO Bertha Gxowa Research Centre, Germiston
- Turkey (Türkiye) (6):
  - Cukurova University Medical Faculty, Adana
  - Gazi University Medical Faculty, Ankara
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Dokuz Eylul University Medicine Faculty, Izmir
  - Erciyes University Medical Faculty, Kayseri
  - Celal Bayar University Medical Faculty, Manisa
- Ukraine (9):
  - CMI Chernivtsi City Children Clinical Hospital, Chernivtsi
  - Regional Children CH Cardiology Department Kharkiv NMU, Kharkiv
  - SI National Research Center of Radiation Medicine of NAMSU, Kyiv
  - USPC of ES EO&T Transplantation of MHU, Kyiv
  - HSEI of Ukraine UMSA, Poltava
  - SSU Division MU Ch of pediatrics, Sumy
  - Vynnitsa Regional Children CH pediatric department № 1 M.I. Pyrogov NMU, Vinnytsia
  - CI Zaporizhzhia City Multibranch Children Hospital #5, Zaporizhzhia
  - CI Zaporizhzhia Regional Clinical Children Hospital of ZRC, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: If the subject was taking antihypertensive medication, the subject was required a 14-day washout. The washout coincided with the Placebo Run-in. The Run-in Period consisted of two visits: Run-in, Day-14 (Visit 2); and Run-in, Day-1 (Visit 3), which only was required for subjects participating in the Ambulatory Blood Pressure Monitoring (ABPM) procedure.
  Participants who were enrolled in the study may have screen failed prior to first dosing with study drug, described above.
Groups:
- Active Comparator: Double Blind Phase: Losartan: 6-week, double-blind (DB), randomized, treatment phase (DB Phase): Starting at Losartan 25/50 and force titrated to 50/100 mg daily at Week 2.
- Experimental: Double-blind: Azilsartan Medoxomil - Low Dose: 6-week, double-blind (DB), randomized, treatment phase (DB Phase): Azilsartan medoxomil Low-dose (AZM-L), 10 mg once daily.
- Experimental: Double-blind: Azilsartan Medoxomil - Medium Dose: 6-week, double-blind (DB), randomized, treatment phase (DB Phase), Azilsartan medoxomil Medium-dose (AZM-M), 20 mg once daily at Week 2.
- Experimental: Double-blind: Azilsartan Medoxomil - High Dose: 6-week, double-blind (DB), randomized, treatment phase (DB Phase): Azilsartan medoxomil High-dose (AZM-H), 40 mg AZM-M
- Placebo Comparator: Withdrawal Phase: PLACEBO: Placebo Arm In the Withdrawal Phase, subjects will be randomized (1:1) to continue taking their previously assigned active treatment or to be switched to placebo.
- Active Comparator: Withdrawal Phase: Losartan 50 mg: Withdrawal Phase, subjects will be randomized (1:1) to continue taking their previously assigned active treatment or to be switched to placebo.
- Active Comparator: WITHDRAWAL Phase: Azilsartan Medoxomil LOW-dose: Experimental Arm in the Withdrawal Phase, subjects will be randomized (1:1) to continue taking their previously assigned active treatment ( Azilsartan medoxomil low dose) that was taken in Double blind OR to be switched to placebo.
- Experimental: WITHDRAWAL Azilsartan Medoxomil - Medium Dose: Experimental Arm in the Withdrawal Phase, subjects will be randomized (1:1) to continue taking their previously assigned active treatment ( Azilsartan medoxomil MEDIUM dose) that was taken in Double blind OR to be switched to placebo.
- Experimental: WITHDRAWAL Azilsartan Medoxomil - High Dose: Experimental Arm in the Withdrawal Phase, subjects will be randomized (1:1) to continue taking their previously assigned active treatment ( Azilsartan medoxomil HIGH dose) that was taken in Double blind OR to be switched to placebo.
- Azilsartan Medoxomil Alone: A subset of subjects taking AZM (10, 20, 40, or 80 mg) alone
- AZM Plus: A subset of subjects taking AZM (10, 20, 40, or 80 mg) plus additional antihypertensives as needed
Period: Double-Blind Phase
Arm/Group | Active Comparator: Double Blind Phase: Losartan | Experimental: Double-blind: Azilsartan Medoxomil - Low Dose | Experimental: Double-blind: Azilsartan Medoxomil - Medium Dose | Experimental: Double-blind: Azilsartan Medoxomil - High Dose | Placebo Comparator: Withdrawal Phase: PLACEBO | Active Comparator: Withdrawal Phase: Losartan 50 mg | Active Comparator: WITHDRAWAL Phase: Azilsartan Medoxomil LOW-dose | Experimental: WITHDRAWAL Azilsartan Medoxomil - Medium Dose | Experimental: WITHDRAWAL Azilsartan Medoxomil - High Dose | Azilsartan Medoxomil Alone | AZM Plus
Started | 53 | 52 | 56 | 54 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 47 | 52 | 53 | 51 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Withdrawal Phase
Arm/Group | Active Comparator: Double Blind Phase: Losartan | Experimental: Double-blind: Azilsartan Medoxomil - Low Dose | Experimental: Double-blind: Azilsartan Medoxomil - Medium Dose | Experimental: Double-blind: Azilsartan Medoxomil - High Dose | Placebo Comparator: Withdrawal Phase: PLACEBO | Active Comparator: Withdrawal Phase: Losartan 50 mg | Active Comparator: WITHDRAWAL Phase: Azilsartan Medoxomil LOW-dose | Experimental: WITHDRAWAL Azilsartan Medoxomil - Medium Dose | Experimental: WITHDRAWAL Azilsartan Medoxomil - High Dose | Azilsartan Medoxomil Alone | AZM Plus
Started | 0 | 0 | 0 | 0 | 103 | 23 | 26 | 26 | 25 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 102 | 22 | 26 | 24 | 23 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 0
Period: Open Label
Arm/Group | Active Comparator: Double Blind Phase: Losartan | Experimental: Double-blind: Azilsartan Medoxomil - Low Dose | Experimental: Double-blind: Azilsartan Medoxomil - Medium Dose | Experimental: Double-blind: Azilsartan Medoxomil - High Dose | Placebo Comparator: Withdrawal Phase: PLACEBO | Active Comparator: Withdrawal Phase: Losartan 50 mg | Active Comparator: WITHDRAWAL Phase: Azilsartan Medoxomil LOW-dose | Experimental: WITHDRAWAL Azilsartan Medoxomil - Medium Dose | Experimental: WITHDRAWAL Azilsartan Medoxomil - High Dose | Azilsartan Medoxomil Alone | AZM Plus
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 156 | 41
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 144 | 40
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 1

BASELINE CHARACTERISTICS:
Population: Demographic Characteristics at Double-Blind Phase
Groups:
- AZM-H: Subjects who received AZM-H
- AZM-M: Subjects who received AZM-M
- AZM-L: Subjects who received AZM-L
- Losartan: Subjects who received Losartan
- Total: Total of all reporting groups
Arm/Group | AZM-H | AZM-M | AZM-L | Losartan | Total
Number analyzed (Participants) | 54 | 56 | 52 | 53 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (2.85) | 13.4 (3.1) | 13.4 (2.92) | 13.2 (3.18) | 13.4 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 40 | 28 | 25 | 118
  Male | 29 | 16 | 24 | 28 | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 14 | 13 | 13 | 55
  White | 37 | 42 | 38 | 38 | 155
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Weight (kg) [Mean (Standard Deviation); unit: kilogram] | 68.97 (24.744) | 66.65 (24.627) | 72.53 (28.556) | 69.00 (26.235) | 69.23 (25.952)

OUTCOME MEASURES:

1. Primary Outcome: Change in Seated Diastolic Blood Pressure Between AZM and Placebo
Description: Change in Seated Diastolic Blood Pressure from Week 6/Final visit of DB Phase to Week 8/Final Visit of the Withdrawal Phase, analysis of study subjects randomized to receiving placebo at Week 6 of treatment versus those who remained on treatment
Time Frame: From Week 6/Final Visit of DB Phase to Week 8/Final Visit of Withdrawal Phase
Population: Analysis of study subjects randomized to receiving placebo at Week 6 of treatment versus those who remained on treatment. The data was pooled for participants who were randomized to receive placebo from Week 6 and pooled for participants who remained receiving AZM treatment from Week 6 to compare the difference in outcome between those who remained on AZM vs. those who changed to placebo. The placebo arms were pooled and the AZM arms were pooled during the DB and Withdrawal phases.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Pooled Placebo: Subjects who received Placebo
- Pooled AZM: Subjects who received AZM
Arm/Group | Pooled Placebo | Pooled AZM
Number analyzed (Participants) | 79 | 77
mmHg | 3.9 (8) | -1.6 (6.69)

2. Secondary Outcome: Change in Trough Seated Systolic Blood Pressure
Description: Change in Trough Seated Systolic Blood Pressure from Week 6 of the Double-Blind Phase to Week 8 of the Withdrawal Phase Between AZM and Placebo, analysis of study subjects randomized to receiving placebo at Week 6 of treatment versus those who remained on treatment
Time Frame: From Week 6/Final Visit of the Double-Blind Phase to Week 8/Final Visit of the Withdrawal Phase
Population: Analysis of study subjects randomized to receiving placebo at Week 6 of treatment versus those who remained on treatment. The data was pooled for participants who were randomized to receive placebo from Week 6 and then pooled for participants who remained receiving AZM treatment from Week 6 to compare the difference in outcome between those who remained on AZM vs. those who changed to placebo. The placebo arms were pooled and the AZM arms were pooled during the DB and Withdrawal phases.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pooled Placebo | Pooled AZM
Number analyzed (Participants) | 79 | 77
mmHg | 4.4 (9.96) | -2.3 (8.72)

3. Secondary Outcome: Change in Mean Arterial Pressure
Description: Change in Mean Arterial Pressure from Week 6 of the Double-Blind Phase to Week 8 of the Withdrawal Phase Between AZM and Placebo, analysis of study subjects randomized to receiving placebo at Week 6 of treatment versus those who remained on treatment
Time Frame: From Week 6 of the Double-Blind Phase to Week 8 of the Withdrawal Phase
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pooled Placebo | Pooled AZM
Number analyzed (Participants) | 79 | 77
mmHg | 4.1 (7.43) | -1.8 (6.63)

ADVERSE EVENTS:
Time Frame: 54 weeks
Description: During the Placebo Run-In period, the pretreatment event/adverse event reported was less than the reporting threshold.
Groups:
- Placebo Run-In: Placebo run-in phase
- Losartan (Double-Blind Phase): Subjects who received Losartan (Double-Blind Phase)
- AZM-L (Double-Blind Phase): Subjects who received AZM-L (Double-Blind Phase)
- AZM-M (Double-Blind Phase): Subjects who received AZM-M (Double-Blind Phase)
- AZM-H (Double-Blind Phase): Subjects who received AZM-H (Double-Blind Phase)
- Placebo (Withdrawal Phase): Subjects who received Placebo (Withdrawal Phase)
- Losartan (Withdrawal Phase): Subjects who received Losartan (Withdrawal Phase)
- AZM-L (Withdrawal Phase): Subjects who received AZM-L (Withdrawal Phase)
- AZM-M (Withdrawal Phase): Subjects who received AZM-M (Withdrawal Phase)
- AZM-H (Withdrawal Phase): Subjects who received AZM-H (Withdrawal Phase)
- Azilsartan Medoxomil Alone: Subjects who receive only AZM
- Azilsartan Medoxomil PLUS: Subjects who receive AZM and any additional antihypertensive therapies
Arm/Group | Placebo Run-In | Losartan (Double-Blind Phase) | AZM-L (Double-Blind Phase) | AZM-M (Double-Blind Phase) | AZM-H (Double-Blind Phase) | Placebo (Withdrawal Phase) | Losartan (Withdrawal Phase) | AZM-L (Withdrawal Phase) | AZM-M (Withdrawal Phase) | AZM-H (Withdrawal Phase) | Azilsartan Medoxomil Alone | Azilsartan Medoxomil PLUS
All-Cause Mortality (participants affected / at risk) | 0/289 | 0/53 | 0/52 | 0/56 | 0/54 | 0/103 | 0/23 | 0/26 | 0/26 | 0/25 | 0/156 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/289 | 2/53 | 1/52 | 1/56 | 0/54 | 0/103 | 0/23 | 1/26 | 0/26 | 0/25 | 7/156 | 2/41
Other Adverse Events (participants affected / at risk) | 0/289 | 6/53 | 5/52 | 6/56 | 5/54 | 6/103 | 0/23 | 4/26 | 0/26 | 0/25 | 11/156 | 32/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Run-In (N=289) | Losartan (Double-Blind Phase) (N=53) | AZM-L (Double-Blind Phase) (N=52) | AZM-M (Double-Blind Phase) (N=56) | AZM-H (Double-Blind Phase) (N=54) | Placebo (Withdrawal Phase) (N=103) | Losartan (Withdrawal Phase) (N=23) | AZM-L (Withdrawal Phase) (N=26) | AZM-M (Withdrawal Phase) (N=26) | AZM-H (Withdrawal Phase) (N=25) | Azilsartan Medoxomil Alone (N=156) | Azilsartan Medoxomil PLUS (N=41)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | NA | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autism spectrum disorder (Psychiatric disorders) | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | NA | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Run-In (N=289) | Losartan (Double-Blind Phase) (N=53) | AZM-L (Double-Blind Phase) (N=52) | AZM-M (Double-Blind Phase) (N=56) | AZM-H (Double-Blind Phase) (N=54) | Placebo (Withdrawal Phase) (N=103) | Losartan (Withdrawal Phase) (N=23) | AZM-L (Withdrawal Phase) (N=26) | AZM-M (Withdrawal Phase) (N=26) | AZM-H (Withdrawal Phase) (N=25) | Azilsartan Medoxomil Alone (N=156) | Azilsartan Medoxomil PLUS (N=41)
Nasopharyngitis (Gastrointestinal disorders) | NA | 3 | 0 | 3 | 2 | 0 | NA | 0 | NA | NA | 0 | 5
Upper respiratory tract infection (Infections and infestations) | NA | 0 | 5 | 0 | 0 | 0 | NA | 2 | NA | NA | 0 | 6
Headache (Nervous system disorders) | NA | 3 | 0 | 3 | 3 | 6 | NA | 2 | NA | NA | 11 | 0
Diarrhoea (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 0 | 0 | NA | 0 | NA | NA | 0 | 3
Gastroenteritis (Infections and infestations) | NA | 0 | 0 | 0 | 0 | 0 | NA | 0 | NA | NA | 0 | 3
Influenza (Infections and infestations) | NA | 0 | 0 | 0 | 0 | 0 | NA | 0 | NA | NA | 0 | 3
Pharyngotonsillitis (Infections and infestations) | NA | 0 | 0 | 0 | 0 | 0 | NA | 0 | NA | NA | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | NA | 0 | 0 | 0 | 0 | 0 | NA | 0 | NA | NA | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 0 | 0 | NA | 0 | NA | NA | 0 | 3
Hypertension (Vascular disorders) | NA | 0 | 0 | 0 | 0 | 0 | NA | 0 | NA | NA | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT02235909/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT02235909/SAP_001.pdf